CLINICAL TRIAL: NCT02765763
Title: Clinical Evaluation of Day and Night Skin Care Creams Supplemented With MediCell Technology (MCT)'s Composition of Defensins and Supportive Molecules
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advanced Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFT Defenage
Record Dates: First submitted 2016-04-11; First posted 2016-05-09 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2016-06

CONDITIONS: Skin Aging; Photoaging of Skin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Sham (Sham Comparator): Null Formula of the Test System
  Interventions: Drug: Null Formula 2-Minute Reveal Masque; Drug: Null Formula 24/7 Barrier Repair Cream; Drug: Null Formula 8-in-1 BioSerum
- Group 2 Treated (Active Comparator): Full Formulas of Test System
  Interventions: Drug: 2-Minute Reveal Masque; Drug: 24/7 Barrier Repair Cream; Drug: 8-in-1 BioSerum

INTERVENTIONS:
Drug: 2-Minute Reveal Masque
  Arms: Group 2 Treated
Drug: 24/7 Barrier Repair Cream
  Arms: Group 2 Treated
Drug: 8-in-1 BioSerum
  Arms: Group 2 Treated
Drug: Null Formula 2-Minute Reveal Masque
  Arms: Group 1 Sham
Drug: Null Formula 24/7 Barrier Repair Cream
  Arms: Group 1 Sham
Drug: Null Formula 8-in-1 BioSerum
  Arms: Group 1 Sham

SUMMARY:
This is a placebo-controlled blinded clinical evaluation of day and night skin care creams supplemented by Medicell Technology's composition of defensins and supportive molecules determine the skin hydration and anti-aging properties of the topical test articles after repeated application to the skin of human subjects.

DETAILED DESCRIPTION:
45 participants will be selected to participate in a placebo-controlled blinded trial comparing the use of the Full Formulas versus the Null Formulas (2 groups). 15 participants will be enrolled at each study site.

Each participant will test the Test System simultaneously as instructed: The Mask one-to-two times a week plus the Cream and the Serum twice daily (morning and evening); the detailed Directions are shown in Exhibit 2. The test System will be applied directly on face, postauricular and neck skin.

All study subjects will also be provided with Skinfo Clean But Not Dry cleanser and EltaMD UV Pure Broad Spectrum Sun Protective Factor (SPF) 47. Subjects will be instructed to wash their face twice daily with the cleanser and apply the sunscreen each morning after application of the Test System.

Both the study subjects and their physicians will be blinded in terms of the treatment group (the Full Formula or the Null Formula).

Subjects will be screening, consented and enrolled according to Good Clinical Practice.

There will be a 1-week washout of any skin care products deemed to be anti-aging. These products would include any using (as a main ingredient) antioxidants, retinol or retinoid, alpha hydroxyl acid, peptides, growth factors. Any other products that are to continue to be used must have been stable for the last 3 months and must be stable for the 12 weeks of the study.

Before beginning treatment, all participants will undergo medical imaging using the VISIA CA, QuantifiCare imaging system or similar non-invasive visual system. Additionally, their skin will be assessed for transepidermal water loss, wrinkle depth and elasticity (non invasive procedures). Optionally, skin will be tested using non-invasive methods for skin color, hydration, sebum content and will be evaluated using ultrasound scanner (DeremaLab Combo or similar).

Skin evaluation will be also performed at baseline, 6 weeks and 12 weeks using the Griffiths scale (2) as well as the skin evaluation scales for pores, superficial wrinkles, deep or muscle induced wrinkles, and skin radiancy, skin turgor, hyperpigmentation, hypopigmentation, erythema and edema in Blinded Evaluator Skin Assessment (Exhibit 3). The evaluation will be performed in person by the blinded investigators.

Subjects will complete a Consumer Questionnaire (Exhibit 4) at baseline, 6 week and 12 week visits.

Weekly phone calls will be made or emails will be sent (+/- 1 week window) to remind subjects to fill out compliance log, use mask, emphasize cream is applied before the serum. Follow-up appointments reminders will also be sent at this time.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Female
* Fitzpatrick Skin Types: I-VI
* Age: 40 - 75 years
* Individuals who will be able to read, understand and give an informed consent relation to the study they are participating in.
* Individuals who will be free of any dermatological or systemic disorder, which in the Principal Investigator's opinion, could interfere with the study results.
* Individuals who will be in general good health and who will complete a preliminary medical history form mandated by the clinic.
* Individuals who will be able to and agree to cooperate with the Investigator and research staff.
* Individuals who will agree to have test products applied in accordance with the protocol and are able to complete the full course of the study.
* Individuals who will agree to have 2 biopsies on the postauricular area if randomly selected.
* Individuals who will agree to not participate in any other study during the entire length of the study and have not participated in a similar study in the past 30 days.

Exclusion Criteria:

* Individuals who are currently taking any medications (topical or systemic) that may mask or interfere with the test results.
* Individuals who have a history of any acute or chronic disease that might interfere with or increase the risk on study participation. (e.g., systemic lupus erythematosus, rheumatoid arthritis, HIV positive).
* Individuals who are diagnosed with chronic skin allergies (atopic dermatitis/eczema) or recently treated skin cancer within the last 12 months.
* Individuals who control their diabetes using insulin.
* Individuals with any history, which in the Investigator's opinion, indicates the potential for harm to the subject or places the validity of the study in jeopardy.
* Individuals who indicate that they are pregnant or are planning to become pregnant or nursing.
* Individuals who have undergone any of the following procedures:

  * Botox within 6 months before enrollment into study and until study completion
  * Injectable filler within 3 months before enrollment into study and until study completion
  * Lasers or tissue tightening devices (ultherapy, radiofrequency, skin tightening, microcurrent or photorejuvenation, photodynamic therapy) within 6 months before enrollment into study and until study completion
  * Sculptra or Bellafill prior to enrollment into the study and until study completion

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for pore size | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for superficial wrinkles | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for deep wrinkles | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for skin radiancy | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for skin turgor | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for hyperpigmentation | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for hypopigmentation | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for erythema | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for edema | Baseline and 12 weeks
Skin Evaluation assessing change from baseline to 12 weeks using Scale from 0 to 4 for scaling and dryness | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy F Taub, MD, Principal Investigator — Advanced Dermatology. LLC
Locations (1):
- Advanced Dermatology, LLC, Lincolnshire, Illinois, United States

IPD SHARING:
Plan to Share IPD: No